CLINICAL TRIAL: NCT02633917
Title: Motor Control Exercises vs Standard Exercises in Patients With Unspecific Low Back Pain
Brief Title: Motor Control Exercises vs Standard Exercises in Unspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Gustavo Plaza Manzano, Director, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CI 10/374
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Low Back Pain
Keywords: Low back pain; Motor control; Joint mobilization
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motor control exercises (Experimental): One group should perform motor control exercises
  Interventions: Behavioral: Motor control exercises
- Standard exercises (Active Comparator): the other group should perform standard physiotherapy exercises
  Interventions: Behavioral: Standard exercises

INTERVENTIONS:
Behavioral: Motor control exercises — exercises to strength the lumbar musculature and control the posture
  Arms: Motor control exercises
Behavioral: Standard exercises — general exercises
  Arms: Standard exercises

SUMMARY:
The purpose of the present study was to evaluate and compare the effects of motor control exercises and standard exercises in the pain, incapacity and medicine intake of subjects with unspecific low-back pain.

DETAILED DESCRIPTION:
Eighty-four subjects with unspecific low-back pain were randomly recruited for the present study. The subjects were randomly allocated into control group (who received one hour of standard physiotherapy exercises every days during ten days) or intervention group (who received one hour of control motor exercises every days during ten days). One month after finishing these ten days, patients should perform a home-based exercises program during two months (control group performed home-based standard physiotherapy exercises; intervention group performed home-based motor control exercises). Pain (visual analogic scale), incapacity index (Roland Morris questionnaire) and medicine intake (diary) were evaluated before the intervention, one month and three months after ending the first ten days of intervention.

ELIGIBILITY:
Inclusion Criteria:

* subjects should be independent to walk
* subjects should have unspecific low back pain during at least the last two months
* subjects should have had at least two recidives of low back pain within the last year

Exclusion Criteria:

* subjects with concomitant pathologies that impede the performance of exercises
* pregnants
* subjects with oncologic pathologies
* subjects with cognitive alterations that impede the understanding of the tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in pain level from baseline at one month and three months after the intervention, measured with a visual analogic scale. | The day before beginning the intervention, one month and three months after the first ten days of intervention
  Visual analogic scale

SECONDARY OUTCOMES:
Change in incapacity index from baseline at one month and three months after the intervention, measured with the Roland Morris questionnaire. | The day before beginning the intervention, one month and three months after the first ten days of intervention
  Roland Morris questionnaire
Change in medication intake from baseline at one month and three months after the intervention, measured with a diary that subjects should complete. | The day before beginning the intervention, one month and three months after the first ten days of intervention
  diary

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Plaza-Manzano, Ph.D, Study Director — Universidad Complutense de Madrid